CLINICAL TRIAL: NCT02056444
Title: Tranexamic Acid Comparison in Hip Replacement (TeACH-R) Trial: Comparative Efficacy of Intravenous Versus Topical Tranexamic Acid for Reducing Blood Loss in Elective Primary Total Hip Arthroplasty.
Brief Title: Efficacy of Intravenous Versus Topical Tranexamic Acid in Primary Total Hip Arthroplasty
Acronym: TeACH-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Douglas Naudie, Consultant Orthopaedic Surgeon, London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TeACH-R Trial
Record Dates: First submitted 2014-02-03; First posted 2014-02-06 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Osteoarthritis
Keywords: Blood conservation; Tranexamic acid; Total hip arthroplasty
MeSH Terms: conditions — Osteoarthritis | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical tranexamic acid (TXA) (Experimental): Single dose 1.5 grams topical TXA infiltrated into the surgical field at time of arthrotomy closure.
  Interventions: Drug: Tranexamic Acid
- Intravenous TXA (Active Comparator): Single 20 mg/kg dose of intravenous TXA administered prior to skin incision.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid
  Other Names: Cyclokapron

SUMMARY:
Bleeding during and after total hip replacement surgery is a primary concern to the surgical and anaesthetic team. Tranexamic acid is a commonly-used drug that helps blood clotting and decreases surgical bleeding. The investigators commonly administer the drug intravenously prior to the procedure. Some patients are unable to receive the drug in this form, because of risks related to blood clotting. The investigators know, from studies in total knee replacement surgery, that the investigators can deliver tranexamic acid directly to the surgical site (topically), with similar benefits and less of the drug absorbed into the bloodstream, resulting in less risk to the patient. The investigators seek to find if similar benefit in terms of reducing blood loss is seen using topical tranexamic acid in hip replacement surgery. The investigators' hypothesis is that the topical form will be equivalent, but not better than the intravenous form for reducing intra- and postoperative bleeding. The investigators also expect to see decreased levels of tranexamic acid in the bloodstream when it is administered topically.

DETAILED DESCRIPTION:
The study randomizes to 2 separate treatment arms: IV administration of tranexamic acid (TXA) at skin incision and topical administration at time of arthrotomy closure. Sample size calculations indicate that 72 study participants in each group would allow for the study sufficient power to detect a clinically relevant change in post-operative hemoglobin levels, in a non-inferiority study design. A double-blind protocol will be implemented, with consent for study participation obtained at the time of the Pre-Admission Clinic appointment.

Randomization will occur as follows: A sealed envelope, appended to the patient chart at the time of the pre-admission clinic appointment, will be provided to the physician at the time of perioperative blood conservation program review. This physician will open the envelope after ensuring that the patient is a candidate to receive TXA. The order will then be placed for either the topical or intravenous form to be sent with the patient to the operating theatre on the day of surgery. The treating surgeon, anaesthesia team, residents and nurses that are in the operating room on the day of surgery will be away of the study participant's randomization, but have been instructed to avoid discussing the administration group to maintain blinding of the patient as best as possible. During the procedure, either the anaesthetist will administer the IV TXA prior to skin incision, or the surgeon will infiltrate, into the surgical wound, the topical TXA at the time of arthrotomy closure. No team members in the operating theatre will be involved in data collection during the post-operative period, and will be instructed not to disseminate any information regarding the route of administration in the electronic or paper chart. Data will then be collected by an independent reviewer not involved in the randomization process, or the procedure itself. In this fashion, the data collectors as well as the participants will be blinded to the intervention. In the immediate postoperative period, the surgical team will be responsible for making clinical decisions, without any influence of the research team. Best efforts will be made to keep the patient unaware of the results of randomization during their in-hospital stay and at the time of any subsequent follow-up visits.

For the intravenous TXA group, administration will follow the current protocol at London Health Sciences Centre (LHSC), where a standard dose of 20 mg/kg will be given to the patient prior to skin incision. For the topical group, a standard dose of 1.5 grams will be given as per the best current evidence in total knee arthroplasty. The latter will be administered at the end of the procedure; the solution will bathe the operative field for 5 minutes during arthrotomy closure, with the final prosthetic components in situ.

Primary outcome measures include differences in postoperative hemoglobin levels and blood transfusion requirements. The investigators routinely measure hemoglobin levels on post-operative days 1 and 2; subsequent measurements are based on suspicion of continued bleeding. Comparison of these levels will be made with levels obtained in the Pre-Admission Clinic appointment to obtain the delta hemoglobin level (delta-Hgb). The lowest measured value during the patient's stay in hospital will be taken as the determinate value. Secondary outcome measures include the number of units of packed red blood cells (pRBC) transfused, as well as the complication rate, both for transfusion-related and procedure-related complications. Packed RBC transfusion as per Health Canada-recommended Clinical Practice Guidelines, at the discretion of the treating surgical team.

The investigators will also measure plasma levels of tranexamic acid intraoperatively, or in the immediate post-operative period, in order to compare the systemic absorption levels with each route of administration. A 5 mL blood sample will be drawn 1 hour after administration. For the intravenous group, this will occur intraoperatively; for the topical route, this will be drawn in PACU. Precise timing of administration and blood sample collection will be marked on the Chart Abstraction Form. 5 mL of blood will be required for this purpose. The specimen will then be sent to to the core laboratory to be cooled and stored until time of centrifugation. Once centrifuged, serum samples will be frozen at -80 degrees Celsius (-80C). Batches of 20 samples will then be sent to St. Michael's Hospital in Toronto, Ontario, for Tandem Mass Spectrometry. This is the only current available method of analysis for serum TEA levels. All 120 participants in this study will have blood levels of TEA measured in this fashion.

ELIGIBILITY:
Inclusion Criteria:

* Primary elective total hip arthroplasty
* Cementless total hip implant system
* Candidate for administration of TEA (as per the LHSC Perioperative Blood Conservation Program Medical Directive titled Preoperative Written Order for Tranexamic Acid in Orthopaedic Surgery)
* Fitness for surgery confirmed after Pre-Admission Clinic appointment
* Consent for transfusion of blood or blood-related products obtained at time of Pre-Admission Clinic appointment.
* Ability to read and understand the English language

Exclusion Criteria:

* Not deemed medically fit for major orthopaedic surgery
* Revision total hip arthroplasty
* Non-elective indication for total hip arthroplasty
* History of thrombotic vascular event (VTE) in the previous 12 months, or requiring lifelong anticoagulation related to previous VTE. VTE is defined as cerebrovascular event (stroke, transient ischemic attack), deep vein thrombosis, and pulmonary embolism
* Consent for transfusion of blood or blood-related products not obtained
* History of developmental hip dysplasia in the operative hip
* History of Legg-Calve-Perthes disease in the operative hip
* Documented allergy to TEA, or to any of its constituent agents
* Unable to participate in scheduled follow-up appointments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2014-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Delta-hemoglobin (ΔHgb) | POD0 to day of discharge (estimated time in hospital 2 to 5 days postop after primary THA)
  (Measured Hgb value closest to operative date) - (lowest Hgb value measured postoperatively in hospital)
Calculated blood loss | POD0 to day of discharge (estimated time in hospital 2 to 5 days postop after primary THA)
  Based on difference between preoperative and postoperative Hgb and hematocrit (Hct) levels.

SECONDARY OUTCOMES:
Venous thromboembolic event (symptomatic deep vein thrombosis or pulmonary embolism) | POD0 to day of discharge (estimated time in hospital 2 to 5 days postop after primary THA); 2 week follow-up; 6 week follow-up; 3 month follow-up.
  Clinically proven symptomatic deep vein thrombosis (DVT) or pulmonary embolism (PE).
Acute coronary syndrome | POD0 to day of discharge (estimated time in hospital 2 to 5 days postop after primary THA); 2 week follow-up; 6 week follow-up; 3 month follow-up.
Cerebrovascular accident (stroke) | POD0 to day of discharge (estimated time in hospital 2 to 5 days postop after primary THA); 2 week follow-up; 6 week follow-up; 3 month follow-up.
Acute kidney injury (AKI) | POD0 to day of discharge (estimated time in hospital 2 to 5 days postop after primary THA); 2 week follow-up; 6 week follow-up; 3 month follow-up.
Pneumonia | POD0 to day of discharge (estimated time in hospital 2 to 5 days postop after primary THA); 2 week follow-up; 6 week follow-up; 3 month follow-up.
  Radiographically-proven pneumonia.
Other systemic illness/infection | POD0 to day of discharge (estimated time in hospital 2 to 5 days postop after primary THA); 2 week follow-up; 6 week follow-up; 3 month follow-up.
  To be specified on the data collection form.
Number of units of packed red blood cell transfused | POD0 to day of discharge (estimated time in hospital 2 to 5 days postop after primary THA)
Hematoma | POD0 to day of discharge (estimated time in hospital 2 to 5 days postop after primary THA); 2 week follow-up; 6 week follow-up; 3 month follow-up.
  Presence of post-operative hematoma near the surgical wound
Length of stay in hospital (days) | POD0 to day of discharge (estimated time in hospital 2 to 5 days postop after primary THA)
  Length of hospital stay after total hip arthroplasty
Systemic serum tranexamic acid (TXA) levels | One hour after administration of TXA
  Blood sample collected one hour after administration, both for the topical and intravenous routes.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas DR Naudie, MD, FRCSC, Principal Investigator — The Joint Replacement Institute at London Health Sciences Centre, University Hospital; James L Howard, MD, MSc, FRCSC, Principal Investigator — The Joint Replacement Institute at London Health Sciences Centre, University Hospital; Richard P Nadeau, BMSc, MD, Principal Investigator — Western University and London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, University Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Ralley FE, Berta D, Binns V, Howard J, Naudie DD. One intraoperative dose of tranexamic Acid for patients having primary hip or knee arthroplasty. Clin Orthop Relat Res. 2010 Jul;468(7):1905-11. doi: 10.1007/s11999-009-1217-8. Epub 2010 Jan 9. PMID 20063079
- [Background] Alshryda S, Mason J, Sarda P, Nargol A, Cooke N, Ahmad H, Tang S, Logishetty R, Vaghela M, McPartlin L, Hungin AP. Topical (intra-articular) tranexamic acid reduces blood loss and transfusion rates following total hip replacement: a randomized controlled trial (TRANX-H). J Bone Joint Surg Am. 2013 Nov 6;95(21):1969-74. doi: 10.2106/JBJS.L.00908. PMID 24196467
- [Background] Imai N, Dohmae Y, Suda K, Miyasaka D, Ito T, Endo N. Tranexamic acid for reduction of blood loss during total hip arthroplasty. J Arthroplasty. 2012 Dec;27(10):1838-43. doi: 10.1016/j.arth.2012.04.024. Epub 2012 Jun 14. PMID 22704229
- [Background] Konig G, Hamlin BR, Waters JH. Topical tranexamic acid reduces blood loss and transfusion rates in total hip and total knee arthroplasty. J Arthroplasty. 2013 Oct;28(9):1473-6. doi: 10.1016/j.arth.2013.06.011. Epub 2013 Jul 23. PMID 23886406